CLINICAL TRIAL: NCT00744835
Title: Atrial Fibrillation Ablation Pilot Study- Study Number AFI-20
Brief Title: Atrial Fibrillation Ablation Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFI-20
Record Dates: First submitted 2008-08-28; First posted 2008-09-01 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Ablation Management
  Interventions: Procedure: Ablation procedure and/or cardioversion

INTERVENTIONS:
Procedure: Ablation procedure and/or cardioversion — Ablation Frontiers Cardiac Ablation System

SUMMARY:
This is a prospective, non-randomized, multicenter, multi-country pilot study to evaluate the safety and effectiveness of the Ablation Frontiers Cardiac Ablation System for the ablative treatment of symptomatic permanent atrial fibrillation.

DETAILED DESCRIPTION:
The study shall be conducted according to ISO 14155. Results of this research study will be used to assess the performance and safety of the System and its components. Data may be combined with similar research at additional sites to create a greater understanding of the endpoints. Up to sixty (60) patients (including "roll-in" or training patients) will be enrolled in a non-randomized study to assess the safety and efficacy of the Ablation Frontiers Cardiac Ablation System. Further studies may be performed to gather additional data regarding the safety and efficacy of the system.

Patients with a history of symptomatic permanent AF, willing and able to sign an informed consent, and meeting all inclusion/exclusion criteria, as identified by the clinical investigator, will be enrolled in the study. Comparative and descriptive statistics will be used to summarize patient outcomes for the specified study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* History of symptomatic permanent atrial fibrillation
* Age between 18 and 70
* Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study

Exclusion Criteria:

* Structural heart disease of clinical significance
* Any prior ablation for atrial fibrillation
* Prior ablation for arrhythmias other than AF within the past three months
* Enrollment in any other ongoing arrhythmia study protocol
* Any ventricular tachyarrhythmias currently being treated where the arrhythmia or the management may interfere with this study
* Active infection or sepsis
* Any history of cerebral vascular disease including stroke or TIAs
* Pregnancy or lactation
* Left atrial thrombus at the time of ablation
* Untreatable allergy to contrast media
* Any diagnosis of AF secondary to electrolyte imbalance, thyroid disease, or any other reversible or non-cardiovascular causes
* History of blood clotting (bleeding or thrombotic) abnormalities
* Known sensitivities to heparin or warfarin
* Severe COPD (identified by an FEV1 < 1)
* Severe comorbidity or poor general physical/mental health that, in the opinion of the investigator, will not allow the patient to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, shortened life expectance, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The acute/chronic safety endpoint is recording of all Severe Adverse Events (device and procedure related) followed for six months. | 6 months

SECONDARY OUTCOMES:
Effectiveness | 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Klinic im Park, Zurich, Switzerland
- United Kingdom (3):
  - Papworth Hospital, Cambridge
  - St. George's University of London, London
  - St. Mary's Hospital, London

REFERENCES:
- See also: Company website — http://www.ablationfrontiers.com